CLINICAL TRIAL: NCT06054932
Title: A Phase I Study of LK101 Monotherapy in Participants With Advanced Solid Tumors to Evaluate the Safety, Tolerability, and Immunogenicity
Brief Title: Safety, Tolerability, and Immunogenicity of LK101 Alone in Participants With Incurable Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Likang Life Science and Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LK101-CT11
Record Dates: First submitted 2023-08-30; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-08

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2weeks-intervals prime dose procedure (Experimental): LK101 will be administered in a prime-boost schedule, which is 4 priming vaccination as 2-weeks-intervals followed by 3 booster vaccinations
  Interventions: Drug: LK101 injection
- 1weeks-intervals prime dose procedure (Experimental): LK101 will be administered in a prime-boost schedule, which is 4 priming vaccination as 1-weeks-intervals followed by 3 booster vaccinations
  Interventions: Drug: LK101 injection

INTERVENTIONS:
Drug: LK101 injection — LK101 administrated Q2W as the prime dose, and Q3W in the boost phase
  Arms: 2weeks-intervals prime dose procedure
Drug: LK101 injection — LK101 administrated QW as the prime dose, and Q3W in the boost phase
  Arms: 1weeks-intervals prime dose procedure

SUMMARY:
This is an open-labeled, single-center phase I study in patients with incurable advanced solid tumors, who failed with all previous standard therapy. The aim is to observe and evaluate the safety, tolerability, and immunogenicity of LK101 injection.

DETAILED DESCRIPTION:
This study is designed to evaluate the safety, tolerability, and immunogenicity of the dose escalation of LK101. We used the traditional "3+3" dose escalation design, Subjects who have been pathologically diagnosed with advanced solid tumors and defined as failing all previous standard therapy. LK101 will be administered in a prime-boost schedule of 4 priming vaccination followed by 3 booster vaccinations. The dose escalation will be conducted in a sequential manner, enrolled patients were initially placed in cohort 1, in which the priming phase is administered at 2-week intervals. And then followed the next cohort 2, where the priming phase is administered at 1-week intervals. Decisions with regard to dose escalation to the next dose level will be made jointly by the investigators and the sponsor. AE data was collected until the 21 days following the last prime dose. safety and immunogenicity will also be used to inform the final dose and schedule. A minimum of 6 patients will be treated at the MTD/RP2D.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent.
* Age 18-75.
* life expectancy ≥3 months.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Subjects with histologically or cytologically confirmed advanced or metastatic solid tumors, unresponsive to standard treatment or for whom no standard treatment is available or appropriate.
* The sequencing of the tumor was qualified.
* Subject must have measurable diseases as per RECIST v1.1 criteria.
* According to the investigator's judgment, venous vascular conditions can meet the needs of apheresis.
* Adequate bone marrow, renal, and hepatic at screening and at Baseline.

Exclusion Criteria:

* Patients who have received therapeutic tumor vaccine products (including peptide vaccine, mRNA vaccine, DC vaccine, etc.).
* Diagnosis of malignant diseases other than study disease within 5 years before screening (except for malignant tumors that can be expected to recover after treatment).
* Patients received systemic antitumor treatment within 2 weeks before the apheresis, or receive research drugs or device therapy.
* Received radiotherapy within 4 weeks prior to screening.
* Toxicity caused by previous treatment did not recover to CTCAE (version 5.0) Grade 1 or below (except hair loss and peripheral neuropathy).
* Patients who have active brain metastases or cancerous meningitis.
* History of significant cardiovascular and cerebrovascular disease occurred in the 6 months prior to screening, Any of the following cardiac criteria:

  * Mean resting corrected QT interval (QTc) > 470 ms;
  * Left ventricular ejection fraction (LVEF) ≤ 50%;
  * American New York heart association (NYHA) heart function ≥ 2 or higher;
  * serious arrhythmia;
  * poorly controlled hypertension;
  * other serious heart diseases;
  * Patients with interstitial pneumonia, except those inactive and do not require hormone therapy disease;
* Any of the following test results are positive: human immunodeficiency virus (HIV) antibody, treponema pallidum antibody, hepatitis C virus (HCV) antibody, hepatitis B virus (HBV) surface antigen (HBsAg), HBV DNA and novel coronavirus nucleic acid.
* Active tuberculosis (TB) during screening.
* Treatment with systemic steroids or other immunosuppressive agents within 14 days prior to screening;
* Vaccination within 4 weeks prior to screening.
* Major injuries and/or surgery =< 4 weeks prior to screening.
* Persons with a history of psychotropic substance abuse and inability to abstain or with a history of mental disorders.
* Pregnant or lactating women.
* Other conditions are regimented at the investigators' discretion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
DLT | Continuously throughout the study until 90 days after Termination of the treatment
  incidence of Dose limited toxicity(DLT),incidence and severity of adverse events (AEs), serious adverse events (SAEs), and immune-related adverse events (irAEs); Clinically significant abnormal changes in laboratory tests and other tests.
AE | Continuously throughout the study until 90 days after Termination of the treatment
  incidence and severity of adverse events
irAE | Continuously throughout the study until 90 days after Termination of the treatment
  incidence and severity of immune-related adverse events
SAE | Continuously throughout the study until 90 days after Termination of the treatment
  incidence and severity of serious adverse events
RP2D | 21 days after the last prime dose
  Recommended phase 2 immune procedure

SECONDARY OUTCOMES:
immunogenicity | 24 months
  neoantigen specific T cell response by ELISpot measurement
ORR | 24 months
  Objective Response Rate (ORR)according to mRECIST 1.1 standard
DoR | 24 months
  Duration of remission
DCR | 24 months
  Disease Control Rate
TTR | 24 months
  Time to remission
TTP | 24 months
  Time to progression
PFS | 24 months
  Progression Free Survival
OS | 24 months
  Overall Survival

OTHER OUTCOMES:
Tumor immune microenvironment before and after treatment | 24 months
  CD8+T cell, PD-1, PD-L1, etc.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Cancer hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality